CLINICAL TRIAL: NCT02126202
Title: Coronary Angioplasty in Octogenarians With Emergent Coronary Syndromes: The Octogenarians Study
Brief Title: Coronary Angioplasty in Octogenarians With Emergent Coronary Syndromes
Acronym: 80+
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Per Albertsson, Head of Cardiology, Sahlgrenska University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 80+
Record Dates: First submitted 2014-01-07; First posted 2014-04-29 (Estimated); Last update posted 2014-04-29 (Estimated); Status verified 2014-01

CONDITIONS: Non-ST Elevation Myocardial Infarction (NSTEMI); Angina, Unstable
Keywords: Elderly; Octogenarians; PCI; Myocardial infarction; NSTEMI; Unstable angina pectoris
MeSH Terms: conditions — Non-ST Elevated Myocardial Infarction; Angina, Unstable; Myocardial Infarction | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conservative therapy (No Intervention): Optimized medical therapy
- Invasive therapy (Experimental): Coronary angiography and revascularization if feasible
  Interventions: Procedure: Coronary angiography and revascularization if feasible

INTERVENTIONS:
Procedure: Coronary angiography and revascularization if feasible — Coronary angiography and revascularization with PCI or CABG (coronary artery bypass grafting) if feasible
  Other Names: Percutaneous coronary intervention (PCI)
  Arms: Invasive therapy

SUMMARY:
A multicenter, randomized clinical trial in elderly patients (over 80 years old) with unstable angina pectoris or Non-ST elevation myocardial infarction (NSTEMI).

A total of 200 patients will be randomized to medical treatment (100 patients) or coronary angiography with revascularization if feasible (100 patients). Information regarding prior history, frailty, clinical presentation, in-hospital events, complications, angina, quality of life and mortality will be collected. Follow up time is 1 year.

ELIGIBILITY:
Inclusion Criteria:

1. >80 years of age
2. Acute coronary syndrome with ischemic symptoms (mainly chest pain) lasting over 10 minutes during the last 72 hours.

   AND at least one of the following:
   1. ST-segment depression on ECG > 1mm
   2. Elevated cardiac troponins
3. Written informed consent before randomization

Exclusion criteria:

1. Percutaneous coronary intervention (PCI) within 30 days prior to randomization
2. Suspected ongoing active internal bleeding
3. ST segment elevation of >1mm in two contiguous leads on ECG
4. Enrollment in another study that has not completed the follow up phase.
5. Known allergy to aspirin or clopidogrel
6. Severe dementia
7. Expected limited 1 year survival due to other disease(s)
8. Unwillingness to participate in the trial or expected problems with compliance

Min Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2009-08; Primary Completion 2015-01 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with major adverse cardiac and cerebral events (the composite of death, myocardial infarction, urgent revascularisation, recurrent hospitalization due to cardiac reason and stroke). | 1 year

SECONDARY OUTCOMES:
Number of participants with major bleeding | 1 month
Number of participants with major adverse cardiac or cerebral event | 1 month
Number of participants with minor bleeding | 1 month
Number of participants with composite of cardiac death or myocardial infarction | 1 year
Change from baseline of participants level of quality of life measured with the SF-36 questionnaire at 12 months | 1 year
Change from baseline of participants level of angina pectoris at 12 months | 12 months
Number of participants dead (all cause mortality) | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Per A Albertsson, PhD, Principal Investigator — Sahlgrenska University Hospital
Locations (1):
- Department of Cardiology, Sahlgrenska University Hospital, Gothenburg, Sweden

REFERENCES:
- [Derived] Hirlekar G, Libungan B, Karlsson T, Back M, Herlitz J, Albertsson P. Percutaneous coronary intervention in the very elderly with NSTE-ACS: the randomized 80+ study. Scand Cardiovasc J. 2020 Oct;54(5):315-321. doi: 10.1080/14017431.2020.1781243. Epub 2020 Jun 26. PMID 32586153
- [Derived] Libungan B, Hirlekar G, Albertsson P. Coronary angioplasty in octogenarians with emergent coronary syndromes: study protocol for a randomized controlled trial. Trials. 2014 Sep 4;15:349. doi: 10.1186/1745-6215-15-349. PMID 25189626